CLINICAL TRIAL: NCT02367768
Title: Long-term Outcome Related Prognostic Factor and Biomarkers of Major Trauma Database Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201410060RINA
Record Dates: First submitted 2015-02-06; First posted 2015-02-20 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Wounds and Injuries
Keywords: trauma blue; major trauma; cohort study; prognostic factor; Healing Time; Post Operative
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CRP, IL-6, cortisol / prolactin / growth hormone
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators were looking for resuscitation management, trauma mechanism, risk factors, and de novo biomarkers related to prognosis and long-term outcome for evaluating trauma patients besides injury severity score (ISS) guiding the traumatologist. The medicare resource could be utilized efficiently along with increasing in the survival and quality of lifer (QoL) in major trauma.

DETAILED DESCRIPTION:
Severe traumatic injury occupied the sixth leading cause of death in Taiwan, especially in young adults. In 2013, there were accidental deaths in every 76 minutes. Not compared with the malignancy, heart disease, cerebrovascular disease, diabetes mellitus, or pneumonia Since 1995, Taiwan replaced a previous patchwork of separate social health insurance funds with one single-payer, National Health Insurance (NHI) scheme that is administered by an agency of the central government's Department of Health. NHI supported the cost of Critical Illness and Injury that numerous patients with major trauma were eligible for preference. However, the national medical cost of trauma care, especially in poly-trauma or major trauma were impressive: the adjusted national inpatient trauma yearly costs were estimated at $37,511,328,659 US dollars; the national insurance cost provided by Bureau of National Health Insurance, Department of Health for trauma was over $20,000,000,000 new Taiwan dollars till 1999 with increasing yearly.

Recently it flashed bulletins nationwide and overseas for catastrophes, such as aircraft accident, wrecks, or underground gas explosions. There was a stirring of interest in life support system for major trauma related rescue from dying. Death to trauma is caused by costly damages on scene, hemorrhage shock or trauma and massive transfusion related acute respiratory distress syndrome (ARDS). Extra-Corporeal Membrane Oxygenation (ECMO) can rescue life from severe cardiopulmonary failure, but coexisting complication as bleeding and coagulopathy restricting the utilization the use in trauma patients. Besides, there were more portable ECMO sets making a debut, especially for air transportation. It act now the medical transferral for trauma patients under ECMO support. The portable ECMO sets launched with possibility, accessibility, and convenience. The issue of life support system utilization, long-term outcome, and medical cost-effectiveness for major trauma patients was worth discussing no matter in National Taiwan University Hospital (NTUH) trauma database or National Health Insurance Research Database (NHIRD).

Immune system alteration was previously considered the mechanism of post-traumatic stress disorder (PTSD). Moreover, an externally experienced traumatic event induces downstream alterations in immune function by reducing methylation.

ELIGIBILITY:
Inclusion criteria:

* age ≧ 20
* willing to join this study and sign the inform consent form by the patients or their contactable families
* ISS score ≧ 16, or meet trauma blue or trauma red criteria
* response to primary resuscitation
* without uncontrolled or major (>1500mL) bleeding.

Exclusion criteria:

* active malignancy before the event of major trauma
* age <20, pregnancy woman, breast-feeding woman, or mental illness
* uncontrolled bleeding with hemoglobin <7g/dL after treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All major trauma (ISS>=16 ) patients sent to NTUH and initiated the trauma team, except children younger than 20 years old, pregnancy woman, breast feeding woman, and those forbidden legally.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-02; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Event related survival | 30 days
  since major trauma event till trauma related death

SECONDARY OUTCOMES:
Functional status | 12 months
  Besides Rehabilitation Complexity Scale (RCS) and Functional Independence Measure (FIM) for traumatic brain injury patients, Glasgow Outcome Scale - Extended (GOS-E) and European Quality of Life Five Dimensions Questionnaire (EQ-5D) are used in concerning longer-term outcome indicators. There are currently no robust measures of patient experience for use in major trauma. Functional status after the major trauma event could be measured using non-clinical outcomes such as return to work, maintenance of education and societal dependency at post injury 3, 6, and 12 months.
over all survival | 2 years
  since major trauma event till death

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Chun Kuo, M.D., Principal Investigator — No.7, Chung San South Road, Taipei City 100, Taiwan (R.O.C.)
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan